CLINICAL TRIAL: NCT06920368
Title: Comparative Study Between the Efficacy of Trans-Septal Quilting Sutures, Nasal Pack and Intranasal Silicon Splint in Endoscopic Septoplasty
Brief Title: Different Techniques for Prevention of Complications After Septoplasty Operation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Yahia Ibrahim Ata, principal invistigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9234837
Record Dates: First submitted 2025-03-20; First posted 2025-04-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Septoplasty
Keywords: complication; quilting; splint; pack; septoplasty; endoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- nasal pack (Active Comparator): pack is put after septoplasty operation for prevention of complication of septoplasty
  Interventions: Procedure: septoplasty with nasal packs
- intra-nasal silicon splint (Active Comparator): intra-nasal silicon splint is put after septoplasty operation for prevention of complication of septoplasty
  Interventions: Procedure: septoplasty with intra-nasal silicon splint
- trans-septal quilting sutures (Active Comparator): trans-septal quilting sutures after septoplasty operation for prevention of complication of septoplasty
  Interventions: Procedure: septoplasty with trans--septal quilting sutures

INTERVENTIONS:
Procedure: septoplasty with nasal packs — Septoplasty to all the patients will be done using general hypotensive anesthesia via cuffed oral endotracheal tube. The patient will be positioned in a slight reverse Trendelenburg position. Local hemostasis will be achieved by injection of lidocaine with epinephrine (1:100000) with placement of topical epinephrine soaked cotton (1:1000) then nasal packs in inserted at the end of operation for prevention of post operative complication
  Arms: nasal pack
Procedure: septoplasty with intra-nasal silicon splint — Septoplasty to all the patients will be done using general hypotensive anesthesia via cuffed oral endotracheal tube. The patient will be positioned in a slight reverse Trendelenburg position. Local hemostasis will be achieved by injection of lidocaine with epinephrine (1:100000) with placement of topical epinephrine soaked cotton (1:1000) then intra-nasal silicon splint is inserted at the end of operation for prevention of post operative complication
  Arms: intra-nasal silicon splint
Procedure: septoplasty with trans--septal quilting sutures — Septoplasty to all the patients will be done using general hypotensive anesthesia via cuffed oral endotracheal tube. The patient will be positioned in a slight reverse Trendelenburg position. Local hemostasis will be achieved by injection of lidocaine with epinephrine (1:100000) with placement of topical epinephrine soaked cotton (1:1000) then trans-septal quilting sutures is done at the end of operation for prevention of post operative complication
  Arms: trans-septal quilting sutures

SUMMARY:
the aim of the study is to compare complication of trans-nasal quilting sutures, nasal pack and intra intranasal silicon splint in endoscopic septoplasty

DETAILED DESCRIPTION:
Septoplasty is the recommended procedure for treating deviated septum and many surgeons are adopting an increasingly conservative approach to septal surgery, such that only the deviated portion of the septum is addressed by the surgery.

The surgical methods utilized in this procedure differ, though the procedure typically involves removal of the deviated cartilage and bony septum that creates a dead space between the mucosal flaps. Although rare, complications such as septal hematoma and consequently abscess formation, adhesions and perforation can occur post-operatively. Three main methods have been employed to prevent such complications. These are intranasal occlusive packing, intranasal silicon splinting, and trans-septal quilting suturing.

However, the totally occlusive nasal packing has many temporary negative effects on the patients' quality of life, which are well studied in the literature. The main disadvantages include: sleep disturbance, patient's discomfort, local pain, headache, dysphagia, breathing difficulty, anxiety and more severe pain on pack removal(6). Bilateral nasal packing may affect the respiratory function due to inadequate oral breathing causing nocturnal hypoxia, which may become more apparent in patients with obstructive sleep apnea or chronic lung diseases. Eustachian tube dysfunction, intranasal infections, toxic shock syndrome, laryngeal or bronchial spasm, myocardial infarction, cerebrovascular accidents has been reported. In addition, the mucosal damage caused by nasal packing may lead to loss of cilia and affects the mucociliary clearance during the healing period.

Intranasal silicone splinting is fast, technically simple and can be used for cartilage support. However, it can cause discomfort in terms of frequent sneezing and epiphora and has a potential risk for bacterial colonization.

The most important advantages of the suture technique include: the non-obliteration of the nasal cavities and the absence of agony associated with pack removal, so it highly decreases patient's discomfort and anxiety related to breathing and pack removal.

the aim of the study is to compare complication of trans-nasal quilting sutures, nasal pack and intra intranasal silicon splint in endoscopic septoplasty

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patient of different ages from 16 to 60 year-old with symptomatic deviated nasal septum

Exclusion Criteria:

* Patient with nasal polyposis or nasal tumors or patients with sinusitis not responding to medical treatment.
* Patient with previous septal operation
* Patient who is planned to do partial inferior turbinectomy or turbinoplasty with septoplasty
* Patients with contraindications for general surgery

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
complication of septoplasty | 1 week, one month and 3 months postoperatively
  endoscopic assessment of post operative recovery and complication
post operative pain | 1 week, 1 month and 3 months postoperatively
  post operative pain will be assessed via Visual Analogue scale ( VAS ) on scale from 0 to 10 as higher scores mean worse outcome.
improvement of nasal symptoms | 1 week, 1 months and 3 months post operatively
  improvement of nasal symptoms will be assessed by using validated Arabic version of NOSE score from 0 to 4 as higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emad Mohamed Shehata, Professor, Principal Investigator — Tanta University Hospitals
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided